CLINICAL TRIAL: NCT03688048
Title: Can Non-drug Antidepressant Treatments Influence the Way the Human Brain Processes Information?
Brief Title: Effects of a Single Dose of Bright Light Treatment on Measures of Affective Information Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government); P1vital Products Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MS IDREC R48997
Record Dates: First submitted 2018-09-18; First posted 2018-09-27 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Bright Light Treatment; Emotion; Facial Expression Recognition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright light treatment (Experimental): Single-dose bright light treatment (1 hour, 10 000 lux)
  Interventions: Device: Bright light treatment lamp
- Sham placebo (Placebo Comparator): Deactivated negative ion generator in conjunction with a plausible cover story
  Interventions: Device: Sham negative ion generator

INTERVENTIONS:
Device: Bright light treatment lamp — Exposure to bright white light (1 hour, 10 000 lux)
  Arms: Bright light treatment
Device: Sham negative ion generator — Placebo treatment with deactivated negative ion generator (1 hour, audible hum, no ions emitted)
  Arms: Sham placebo

SUMMARY:
This study aims to investigate the effects of a single session of bright light treatment (BLT) on emotional information processing in healthy volunteers. We hypothesised that BLT can acutely push the processing of emotional information towards a prioritisation of positive (relative to negative) input. To test this hypothesis, healthy volunteers were randomly allocated to receive either bright light treatment or sham-placebo treatment and study participants as well as investigators were blind as to which treatment was used. After treatment, all participants underwent testing with the Oxford Emotional Test Battery, an established set of psychological tasks that allow to assess how emotional information is processed.

DETAILED DESCRIPTION:
Background:

Bright light treatment (BLT) is an efficacious treatment for depressive disorders but the causal mechanisms by which it exerts its clinical effects are largely unknown. According to the cognitive neuropsychological model of antidepressant treatment action, one way by which antidepressant treatments lead to clinical effects is by acutely inducing a relatively increased preferential processing of positive (as compared to negative) emotional stimuli. Whether BLT has the potential to induce such positive biases is not known to date.

Aim of study:

To investigate the influence of single-dose BLT on emotion-related information processing in healthy volunteers.

Methods:

Using a double-blind, parallel-group design, fifty healthy volunteers (male and female) were randomly allocated to a single session (60 minutes) of treatment with either bright light (10 000 lux) or a credible placebo-sham condition (deactivated negative ion generator). After treatment, all participants underwent testing with the Oxford Emotional Test Battery, an established battery of behavioural tasks that allow to assess emotional information processing in multiple cognitive domains. This battery consists of a facial expression recognition task, an emotional categorization task, an emotional dot probe task, an emotional recall task and an emotional recognition task. Before and after treatment, subjective state was assessed using different questionnaires.

Hypotheses:

Our working hypothesis, in line with the cognitive neuropsychological model of antidepressant treatment action, is that one-time BLT can induce biases towards positive stimuli in multiple cognitive domains and this bias will be present even in the absence of observable changes in subjective state.

Implications of the study:

This study will show whether a single dose of BLT can influence emotion-related information processing in a similar way as previously observed for antidepressant drugs. If this is the case, then the clinical effects of BLT could be explained through its acute effects on emotional processing. On a broader level, the results of this study will also add to our understanding of any potential effects that acute exposure to bright light (e.g. sunlight) could have on the healthy human mind.

ELIGIBILITY:
Entry criteria:

1. Female or male
2. Age: 18 to 65 years
3. Good general health
4. Competency to give informed consent

Exclusion criteria:

1. Any current or past psychiatric disorder
2. Any first-degree relative with a diagnosis of schizophrenia-spectrum or other psychotic disorder, bipolar disorder, or depressive disorder
3. Any severe medical condition not stabilized at the time of the experiment (e.g. asthma, heart disease)
4. Any condition which precludes treatment with bright light (e.g. retinal disorder, intake of photo-sensitizing medication)
5. Any current or past physical illness that has the potential to significantly affect mental functioning (e.g. stroke, Parkinson's disease)
6. Pregnant, lactating, or sexually active women who do not use any medically accepted method of contraception
7. Any history of seizures or any condition with the potential to manifest with seizures (e.g. epilepsy)
8. Diagnosis of diabetes (because of potential risk of retinal disorder)
9. Current intake of medication that has a significant potential to affect mental functioning, or intake of such medication in the previous 3 months (e.g. antidepressants, neuroleptics, tranquilizers)
10. Any intake of recreational drugs in the last 3 months before the experiment
11. Excessive alcohol consumption up to three days before the experiment
12. Previous use of bright light treatment or negative ion treatment
13. Participant usually (more than 5 days a week) gets up later than 10.00 a.m.
14. Necessity to wear tinted glasses
15. Any kind of sun exposure in the last month that is unusually high for local conditions (e.g. beach vacation, skiing holidays)
16. The researchers decide to exclude a participant for any other reason (because participation could be harmful to a participant, or a participant can't properly interact with the researchers or could bias the study results)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Performance in a facial expression recognition task | Completed within 2 hours after treatment
  Participants are presented with individual pictures of facial expressions of emotions. Each presented face displays one of six basic emotions (anger, disgust, fear, happiness, sadness, or surprise). Each emotional expression is presented at different levels of intensity which have been created by combining shape and texture features of the two extremes "neutral" (0%) and "full prototypical emotion" (100%) to varying degrees. Examples of neutral facial expressions are presented as well. Participants are instructed to correctly classify each facial expression as angry, disgusted, fearful, happy, sad, surprised or neutral both as quickly and as accurately as possible. Responses are made by pushing one out of seven labelled keys on a response box. Hit rates, false alarm rates, and reaction times for correct classifications are measured separately for each emotion.

SECONDARY OUTCOMES:
Performance in an emotional categorisation task | Completed within 2 hours after treatment
  Participants are presented with positive and negative personality descriptors and are asked to classify the valence of each word. These words describe either extremely agreeable/positive characteristics (e.g. "cheerful", "honest", "optimistic") or extremely disagreeable/negative characteristics (e.g. "domineering", "untidy", "hostile") and are presented individually in the centre of the screen. Participants are instructed to imagine themselves overhearing someone describing them with each of the words and to indicate as quickly and accurately as possible whether they would like or dislike to be described with each of the words. Responses are made by pressing a correspondingly labelled key on a button box. Reaction times for correct classifications are measured separately for positive and negative words.
Performance in an emotional faces dot probe task | Completed within 2 hours after treatment
  Pictures of positive and negative emotional stimuli (happy and fearful facial expressions) are presented individually together with a matched neutral stimulus (neutral face). On each trial, one stimulus is shown above and the other below a central fixation point. Subsequently, a probe appears behind one of the stimuli and participants have to correctly classify the probe as quickly and as accurately as possible. Stimuli can be masked (i.e. presented very briefly and followed by a jumbled face) or unmasked (i.e. presented for a longer period without a subsequent masking stimulus). Reaction times for correct responses are recorded and vigilance scores are calculated for masked and unmasked positive and negative stimuli by subtracting reaction time data from trials when the probe appeared in the same position as the emotional stimulus (congruent trials) from trials when the probe appeared in the opposite position to the emotional stimulus (incongruent trials).
Performance in an emotional recall task | Completed within 2 hours after treatment
  Following a delay period after the emotional categorization task (about 15 min), emotional recall memory is assessed. Participants are asked to recall and write down as many words as possible from the emotional categorization task. Numbers of correctly and incorrectly recalled positive and negative words are measured.
Performance in an emotional recognition task | Completed within 2 hours after treatment
  Following the emotional recall task, emotional recognition memory is assessed by presenting participants with the original personality descriptors plus an equal number of matched distractor words (50% positive, 50% negative). Participants are asked to indicate for each word as accurately and as quickly as possible whether they recognise it from the emotional categorization task. Numbers of correctly and incorrectly recognised items as well as reaction times for correct recognitions are measured separately for positive and negative words.

OTHER OUTCOMES:
Change in subjective mood and energy | Completed within 2 hours after treatment
  Zersen's Befindlichkeits-Skala. Standard questionnaire for subjectively felt mood and energy levels. Total score ranging from 0 to 112. Subscores: Mood (ranging from 0 to 94) and Energy (ranging from 0 to 18). Sum of subscores for mood and energy provide total score. Higher scores represent worse subjective mood and energy.
Change in positive and negative affect | Completed within 2 hours after treatment
  Positive and Negative Affect Schedule; standard questionnaire for subjectively felt positive and negative affect. Two scores: (1) Positive score: ranging from 10 to 50 (higher score representing greater extent of positive affect). (2) Negative score: ranging from 10 to 50 (higher score representing greater extent of negative affect).
Change in subjective anxiety | Completed within 2 hours after treatment
  State-Trait Anxiety Inventory; standard questionnaire for subjectively felt anxiety. Two scores: (1) State anxiety: ranging from 20 to 80 (higher scores indicating higher state anxiety levels). (2) Trait Anxiety: ranging from 20 to 80 (higher scores indicating higher trait anxiety levels).
Change in subjective state | Completed within 2 hours after treatment
  Visual Analogue Scales of different subjective states (anxious, alert, happy, sad, angry, disgusted, afraid); Minimum = 0 mm ("Not at all") , Maximum = 96 mm ("Extremely"); greater scores represent greater extent of felt emotions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lam RW, Levitt AJ, Levitan RD, Michalak EE, Cheung AH, Morehouse R, Ramasubbu R, Yatham LN, Tam EM. Efficacy of Bright Light Treatment, Fluoxetine, and the Combination in Patients With Nonseasonal Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jan;73(1):56-63. doi: 10.1001/jamapsychiatry.2015.2235. PMID 26580307
- [Background] Golden RN, Gaynes BN, Ekstrom RD, Hamer RM, Jacobsen FM, Suppes T, Wisner KL, Nemeroff CB. The efficacy of light therapy in the treatment of mood disorders: a review and meta-analysis of the evidence. Am J Psychiatry. 2005 Apr;162(4):656-62. doi: 10.1176/appi.ajp.162.4.656. PMID 15800134
- [Background] Harmer CJ, Goodwin GM, Cowen PJ. Why do antidepressants take so long to work? A cognitive neuropsychological model of antidepressant drug action. Br J Psychiatry. 2009 Aug;195(2):102-8. doi: 10.1192/bjp.bp.108.051193. PMID 19648538
- [Background] Roiser JP, Elliott R, Sahakian BJ. Cognitive mechanisms of treatment in depression. Neuropsychopharmacology. 2012 Jan;37(1):117-36. doi: 10.1038/npp.2011.183. Epub 2011 Oct 5. PMID 21976044